CLINICAL TRIAL: NCT06861764
Title: The Relationship Between Preoperative Anxiety and Postoperative Delirium in Elderly Chinese Patients: a Multicenter Prospective Cohort
Brief Title: The Relationship Between Preoperative Anxiety and Postoperative Delirium in Elderly Chinese Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other); Peking University First Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Xiangya Hospital of Central South University (Other); Beijing Anzhen Hospital (Other); Central South University (Other); Peking University People's Hospital (Other); Zhejiang University (Other); Fudan University (Other); Sun Yat-sen University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); China-Japan Friendship Hospital (Other); The Affiliated Hospital Of Guizhou Medical University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Taihe Hospital (Other); Zhejiang Provincial People's Hospital (Other); Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-PA-PD
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Cohort Studies
Keywords: preoperative anxiety; Aged; postoperative delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Preoperative anxiety: According to the GAD-7 scale, the population was defined as the Preoperative anxiety group
- Non-preoperative anxiety: According to the GAD-7 scale, the population was defined as the Non-preoperative anxiety group

SUMMARY:
This study is a retrospective analysis of a large-scale multicentre prospective cohort study that investigates the the relationship between Preoperative Anxiety and Postoperative Delirium in Elderly Chinese Patients: a Multicenter Prospective Cohort

DETAILED DESCRIPTION:
This is a retrospective cohort study using prospective data from a multicenter database. 8000 elderly patients undergoing elective non-cardiac or non-neurosurgical surgery were included in this study. The Generalized Anxiety Disorder Scale (GAD-7) was used to measure preoperative anxiety symptoms. The confusion assessment method (3D-CAM) was used to assess postoperative delirium in elderly patients undergoing non-cardiac surgery. If the patient is discharged, follow up by phone or email. Binary logistic regression analysis and propensity score matching (PSM) and subgroup analysis were used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* elderly patients (age ≥ 65 years)
* non-cardiac surgery, non-neurosurgical surgery

Exclusion Criteria:

* History of neurological or psychiatric disorders or use of neuropsychiatric drugs;
* Impaired cognitive function or inability to cooperate with preoperative follow-up;
* Sent to ICU after surgery;
* Deletional delirium outcome;
* Baseline missing >5%

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly patients (aged ≥ 65 years) who completed the anxiety assessment after the elective noncardiac, non-neurosurgical surgery were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium | within 7 days after surgery
  The incidence of postoperative delirium was assessed by a 3-minute diagnostic interview in the surgical ward (3D-CAM).

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided